CLINICAL TRIAL: NCT01387165
Title: A Multi-center, Epidemiologic Survey to Describe the Current Medical Practice of General Practitioners Treating Subjects With Type 2 Diabetes Mellitus in Latin America
Brief Title: Epidemiologic Survey to Describe the Current Medical Practice of General Practitioners Treating Subjects With Type 2 Diabetes Mellitus in Latina
Acronym: DEAL
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 105407
Record Dates: First submitted 2011-04-14; First posted 2011-07-04 (Estimated); Last update posted 2017-06-08 (Actual); Status verified 2017-05

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Latin America; diabetes complications; patient compliance; Diabetes mellitus, type 2; health services accessibility
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Complications; Patient Compliance | interventions — Therapeutics

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients: males and females between 18 and 75 years of age who been diagnosed with T2DM as defined by the American Diabetes Association
  Interventions: Drug: Treatment

INTERVENTIONS:
Drug: Treatment — were receiving an oral hypoglycemic agent (OHA) or insulin

SUMMARY:
The DEAL (Diabetes En America Latina) study was a multicenter, cross-sectional, epidemiological, questionnaire based study carried out between October 2004 and October 2005 in 9 Latin American countries.

DETAILED DESCRIPTION:
The DEAL (Diabetes En America Latina) study was a multicenter, cross-sectional, epidemiological, questionnaire based study carried out between October 2004 and October 2005 in 9 Latin American countries. General practitioners (GP) from private settings were selected for participation in the study if they were in full time active clinical practice (three or more days per week and treating at least 100 patients per week), had been practicing for at least two years and were seeing at least five type 2 diabetes mellitus (T2DM) patients per week. Over a period of two weeks after receipt of study questionnaires, GPs were required to review the charts of the first 10 (+/- 2) consecutive diabetic patients to visit the clinic and to provide information about their treatment in accordance with the supplied questionnaire.

Patients were eligible for inclusion in the study if they were males or females aged 18-75 with Type II Diabetes Mellitus - T2DM - (defined by the criteria of the American Diabetes Association (12)), were receiving an oral hypoglycemic agent (OHA) or insulin and had given written informed consent, where required. Measurement of glycosylated hemoglobin (HbA1c) performed at the diagnosis and within the previous three months was collected; if the measure was not available for the period, the sponsor supported the laboratory test when necessary, according to the physician's judgment of the patient's need.

Demographic data were collected including information regarding the patient's lifestyle. The most recent fasting blood glucose, lipid level and blood pressure measurements were recorded along with the existence of diabetes related complications such as dyslipidemia, hypertension, macrovascular diseases, eye disorders, kidney disorders, erectile dysfunction and diabetic neuropathy. Antidiabetic medication and/or insulin therapy and therapy for prevention of macrovascular events were also recorded. Information was collected on visits to specialists, challenges to managing the patient's T2DM and on future plans for management. No explanations or clarifications related to the questions were provided and the physicians answered them based on their own understanding. Instructions on how to answer the questionnaire were provided to maximize the validation of the questionnaires.

Descriptive statistical analysis was performed on all variables. Multivariate logistic regression analyses were performed to test the possibility of association between the outcome measures and duration of disease. The independent variables were age, gender, BMI (body-mass index) category, current prescription, drug insurance coverage, glycemic management, lifestyle, number of co-morbidities and compliance to recommendations/therapy. All statistical analyses were conducted using SAS software. A p value <0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Males and females 18-75 years of age, inclusive,
* Males and females with T2DM, as defined by the criteria of the American Diabetes Association (2003),
* Males and females under oral anti-diabetics (OAD) or insulin treatment for diabetes and
* Males and females that have given written informed consent.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Males and females 18-75 years of age, inclusive, with T2DM, as defined by the criteria of the American Diabetes Association (2003), under oral anti-diabetics (OAD) or insulin treatment for diabetes and that have given written informed consent.
  The total number of patients planned for this study was up to 6,000 patients: Mexico - 1,500, Argentina - 1,000, Brazil - 1,500, CariCam - 1,100 (Colombia, Costa Rica, Ecuador, Guatemala, Honduras, Peru, Dominican Republic and Venezuela) and Chile - 500.
Sampling Method: Probability Sample
Enrollment: 3592 (Actual)
Dates: Start 2004-10; Primary Completion 2005-10 (Actual); Study Completion 2005-10 (Actual)

PRIMARY OUTCOMES:
The achievement of the planned completed number of questionnaires. | up to 1 year

SECONDARY OUTCOMES:
Changes in glycemic parameters in accordance with the historical information provided by the GPs and her/his judgement of control based on that information. | up to 1 year
Proportion of subjects who respond to any given treatment applied through the level of HbA1c responders (defined as subjects who have achieved HbA1c <7%) | up to 1 year
Assessment of total cholesterol | up to 1 year
Assessment of free fatty acids | up to 1 year
Assessment of high-density lipoprotein | up to 1 year
Assessment low-density lipoprotein | up to 1 year
Assessment of triglycerides | up to 1 year
Assessment of LDL relative flotation | up to 1 year
Assessment of total cholesterol/HDL ratio | up to 1 year
Assessment of LDL/HDL ratio | up to 1 year
Assessment of fasting blood glucose | up to 1 year

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline

REFERENCES:
- See also: Control of type 2 diabetes mellitus among general practitioners in private practice in nine countries of Latin America — http://www.scielosp.org/pdf/rpsp/v22n1/a02v22n1.pdf